CLINICAL TRIAL: NCT00265850
Title: A Phase III Trial of Irinotecan / 5-FU / Leucovorin or Oxaliplatin / 5-FU/ Leucovorin With Bevacizumab, or Cetuximab (C225), or With the Combination of Bevacizumab and Cetuximab for Patients With Untreated Metastatic Adenocarcinoma of the Colon or Rectum
Brief Title: Cetuximab and/or Bevacizumab Combined With Combination Chemotherapy in Treating Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); SWOG Cancer Research Network (Network); Bristol-Myers Squibb (Industry); Aptuit (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB 80405; U10CA037447 (NIH); CDR0000455161 (Other: Physician Data Query); NCI-2009-00434 (Registry Identifier: NCI Clinical Trial Reporting Program Office)
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Results first posted 2017-04-26 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-04

CONDITIONS: Colorectal Cancer
Keywords: recurrent colon cancer; stage III colon cancer; stage III rectal cancer; stage IV colon cancer; recurrent rectal cancer; stage IV rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab; Cetuximab; Folfox protocol; Oxaliplatin; Leucovorin; Fluorouracil; IFL protocol; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A: FOLFOX or FOLFIRI + bevacizumab (Active Comparator): Patients receive bevacizumab 5 mg/kg IV every two weeks and then receive either FOLFOX or FOLFIRI every two weeks as described in the intervention section. One cycle is defined as 8 weeks of treatment. Treatment continues until disease progression, unacceptable toxicity or surgery with curative intent as planned.
  Interventions: Biological: bevacizumab; Drug: FOLFOX or; Drug: FOLFIRI
- Arm B: FOLFOX or FOLFIRI + cetuximab (Experimental): Patients receive cetuximab 400mg/m^2 IV over 2 hours on the first day of treatment, then 250 mg/m^2 IV over 1 hour weekly thereafter. Patients also receive either FOLFOX or FOLFIRI every two weeks as described in the intervention section. One cycle is defined as 8 weeks of treatment. Treatment continues until disease progression, unacceptable toxicity or surgery with curative intent as planned.
  Interventions: Biological: cetuximab; Drug: FOLFOX or; Drug: FOLFIRI
- Arm C: FOLFOX or FOLFIRI + cetuximab + bevacizumab (Experimental): Patients receive cetuximab 400mg/m^2 IV over 2 hours on the first day of treatment, then 250 mg/m^2 IV over 1 hour weekly thereafter. Also, patients receive bevacizumab 5 mg/kg IV every two weeks and then receive either FOLFOX or FOLFIRI every two weeks as described in the intervention section. One cycle is defined as 8 weeks of treatment. Treatment continues until disease progression, unacceptable toxicity or surgery with curative intent as planned.
  Interventions: Biological: bevacizumab; Biological: cetuximab; Drug: FOLFOX or; Drug: FOLFIRI

INTERVENTIONS:
Biological: bevacizumab — Given IV
  Arms: Arm A: FOLFOX or FOLFIRI + bevacizumab; Arm C: FOLFOX or FOLFIRI + cetuximab + bevacizumab
Biological: cetuximab — Given IV
  Arms: Arm B: FOLFOX or FOLFIRI + cetuximab; Arm C: FOLFOX or FOLFIRI + cetuximab + bevacizumab
Drug: FOLFOX or — Patients receive oxaliplatin 85 mg/m^2 IV infused over two hours followed by leucovorin 400 mg/m^2 IV over 2 hours followed by 5-FU 400 mg/m^2 IV bolus, then 2400 mg/m^2 continuous IV infusion over 46-48 hours
  Other Names: Eloxatin (oxaliplatin), leucovorin (folinic acid) and 5-Fluorouracil (5-FU)
Drug: FOLFIRI — Patients receive irinotecan 180 mg/m^2 IV infused over 90 minutes followed by leucovorin 400 mg/m^2 IV over 2 hours followed by 5-FU 400 mg/m^2 IV bolus following leucovorin then 2400 mg/m^2 continuous IV infusion over 46-48 hours.
  Other Names: CPT-11 (irinotecan), leucovorin (folinic acid), and 5-Fluorouracil (5-FU)

SUMMARY:
PURPOSE: This randomized phase III trial is studying cetuximab and/or bevacizumab when given together with combination chemotherapy to compare how well they work in treating patients with metastatic colorectal cancer.

RATIONALE: Monoclonal antibodies, such as cetuximab and bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Cetuximab may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Drugs used in chemotherapy, such as fluorouracil, leucovorin, oxaliplatin, and irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving monoclonal antibodies together with combination chemotherapy may kill more tumor cells. It is not yet known whether combination chemotherapy is more effective with cetuximab and/or bevacizumab in treating patients with colorectal cancer.

DETAILED DESCRIPTION:
OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to physician-selected chemotherapy (FOLFOX or FOLFIRI), prior adjuvant chemotherapy (yes vs no), and prior pelvic radiotherapy (yes vs no). Patients were randomized to 1 of 3 treatment arms.

Primary Objective:

* To determine if the addition of cetuximab to FOLFIRI or FOLFOX chemotherapy prolongs survival compared to FOLFIRI or FOLFOX with bevacizumab in patients with untreated, advanced or metastatic colorectal cancer who have K-ras wild type tumors.

Secondary Objectives:

* To evaluate response, progression-free survival (PFS), time to treatment failure (TTF), and duration of response (DR) among patients with unresectable advanced metastatic colon cancer treated with bevacizumab or cetuximab in addition to chemotherapy with FOLFIRI or FOLFOX
* To evaluate toxicity and, in particular, 60-day mortality among patients with unresectable advanced metastatic colon cancer treated with bevacizumab or cetuximab in addition to chemotherapy with FOLFIRI or FOLFOX
* To describe patients with unresectable locally advanced or metastatic colorectal cancer rendered "resectable" with chemotherapy

There are premedication guidelines that were established for patients assigned to receive cetuximab. All patients must be premedicated with diphenhydramine hydrochloride 50 mg (or a similar agent) IV prior to the first dose of cetuximab in an effort to prevent an infusion or hypersensitivity reaction. Premedication is also recommended prior to subsequent doses, but at the investigator's discretion the dose of diphenhydramine (or a similar agent) may be reduced. Pretreatment with acetaminophen may also be used.

There are bevacizumab administration instructions for patients for whom surgery is being contemplated or required. For patients for whom elective surgery is contemplated, bevacizumab is to be discontinued for at least 8 weeks prior to surgery. Bevacizumab may be resumed after at least 4 weeks following surgery. Patients who undergo complete resection of metastatic disease will discontinue protocol therapy and may receive further treatment at the treating physician's discretion. For patients for whom non-elective surgery is required, hold bevacizumab as long as possible prior to surgery and for at least 6 weeks following surgery.

Patients received a minimum of two cycles of therapy. Patients were allowed to receive ancillary therapy per protocol. Treatment continued until disease progression, unacceptable toxicity, or surgery with curative intent as planned. After completion of study treatment, patients are followed up to 5 years.

ELIGIBILITY:
1. Locally Advanced or Metastatic Colorectal Cancer

   1. Eligible patients must have histologically or cytologically documented adenocarcinoma of the colon or rectum. Patients must have either locally advanced (unresectable) or metastatic disease. Patients with resected primary tumors who have documented metastases are eligible. Documentation of residual disease by CT scan or surgeon's notes is required for all patients, and histologic confirmation of metastases is strongly encouraged.
   2. Patients with a history of colorectal cancer treatment by surgical resection who develop radiological or clinical evidence of metastatic cancer do not require separate histological or cytological confirmation of metastatic disease unless:

      * Either an interval of greater than five years has elapsed between the primary surgery and the development of metastatic disease or
      * The primary cancer was stage I. Clinicians should consider biopsy of lesions to establish the diagnosis of metastatic colorectal cancer in each case if there is substantial clinical ambiguity regarding the nature or source of apparent metastases.
   3. At the time of randomization, the intent of this treatment must be indicated palliative or neoadjuvant chemotherapy with the potential for resection of all sites of metastatic disease.
2. Only patients with a wildtype K-ras gene as determined by the laboratory at the SWOG Solid Tumor Repository or by a local CLIA-certified laboratory are eligible. Patients with a mutation in the K-ras gene are ineligible. All patients must have available for analysis of K-ras status at least one H and E slide and one paraffin block of the previously resected primary colorectal tumor and/or a tumor deposit. For patients registered and randomized based on local CLIA-certified laboratory results, SWOG analysis will be confirmatory only.
3. Prior Treatment

   1. No prior systemic treatment for advanced or metastatic colorectal cancer is allowed. Prior regional chemotherapy (eg, hepatic arterial infusion) is also not allowed.

      * Patients may have received prior adjuvant chemotherapy that included fluorouracil alone or in combination with fluorouracil and oxaliplatin or irinotecan (no more than 6 months); or radiation with radiosensitizing chemotherapy.
      * The last course of adjuvant chemotherapy must have concluded > 12 months prior to colorectal cancer recurrence.
      * Patients may have received neoadjuvant chemo-radiation with capecitabine or 5-fluorouracil.
      * Patients may not have received itraconazole or ketoconazole less than 4 weeks prior to randomization.
      * No prior exposure to any tyrosine kinase inhibitors or other agents (including protein products, monoclonal antibodies, antisense, etc.) that target VEGF or EGF receptors is allowed.
      * No prior treatment with bevacizumab or cetuximab.
   2. Patients may not have had prior radiotherapy to greater than 25% of bone marrow.

      (Standard adjuvant rectal cancer chemoradiation will not exclude patient from protocol entry.) Radiation must have concluded ≥ 4 weeks prior to randomization.
   3. Patients should have completed any major surgery ≥ 4 weeks from randomization. Patients must have completed any minor surgery ≥ 2 weeks prior to randomization. Patients must have fully recovered from the procedure. (Insertion of a vascular access device is not considered major or minor surgery.)
4. No previous or concurrent malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for five years.
5. For patients who are to receive FOLFIRI: No evidence of Gilbert's Syndrome or of homozygosity for the UGT1A1*28 allele.

   1. Patients with Gilbert's Syndrome may have a greater risk of irinotecan toxicity due to the abnormal glucuronidation of SN-38. Evidence of Gilbert's Syndrome would include a prior finding of an isolated elevation of indirect bilirubin.
   2. UGT1A1 genotyping is not required on this study. However, patients known to be homozygous for the UGT1A1*28 allele are not to receive FOLFIRI for this study. Patients with Gilbert's Syndrome or who are found to be homozygous for the UGT1A1 allele who will receive FOLFOX are eligible.
6. No sensory peripheral neuropathy of ≥ grade 2 at baseline for patients who are to receive FOLFOX.
7. No known central nervous system metastases or carcinomatous meningitis.
8. No interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung.
9. No pleural effusion or ascites that causes ≥ grade 2 dyspnea.
10. No predisposing colonic or small bowel disorders in which the symptoms are uncontrolled as indicated by baseline pattern of > 3 watery or soft stools daily in patients without a colostomy or ileostomy. Patients with a colostomy or ileostomy may entered at investigator discretion.
11. Patients must not have an uncontrolled seizure disorder, or active neurological disease.
12. No current congestive heart failure (New York Heart Association Class II, III or IV)
13. Patients with history of hypertension must be well controlled ( < 160/90) on a regimen of anti-hypertensive therapy.
14. Patients on full-dose anticoagulation (eg, warfarin) are eligible provided that both of the following criteria are met:

    1. The patient has an in-range INR (usually between 2 and 3) on a stable dose of oral anticoagulant or be on a stable dose of low molecular weight heparin.
    2. The patient has no active bleeding or pathological condition that carries a high risk of bleeding (eg, tumor involving major vessels or known varices).
15. Patients receiving anti-platelet agents are eligible. In addition, patients who are on daily prophylactic aspirin or anticoagulation for atrial fibrillation are eligible.
16. No significant history of bleeding events or GI perforation:

    1. Patients with a history of significant bleeding episodes (eg, hemoptysis, upper or lower GI bleeding ) within 6 months of randomization are not eligible unless the source of bleeding has been resected.
    2. Patients with a history of GI perforation within 12 months of randomization are not eligible.
17. No arterial thrombotic events within 6 months before randomization, including transient ischemic attack (TIA), cerebrovascular accident (CVA), unstable angina or angina requiring surgical or medical intervention in the past 6 months, or myocardial infarction (MI). Patients with clinically significantly peripheral artery disease (eg, claudication on less than one block) or any other arterial thrombotic event are also ineligible.
18. No serious or non-healing wound, ulcer or bone fracture
19. Patients with known hypersensitivity to Chinese hamster ovary cell products or to recombinant human or murine antibodies are not eligible.
20. Non-pregnant and not nursing:

    1. Women of child bearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to randomization.
    2. DNA alkylating agents are known to be teratogenic, and the effects of irinotecan, oxaliplatin, 5-FU, bevacizumab, and cetuximab on a developing fetus at the recommended therapeutic doses are unknown.
    3. Women of child-bearing potential include any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal.
    4. Postmenopausal is defined as amenorrhea ≥ 12 consecutive months or women on hormone replacement therapy (HRT) with documented serum follicle stimulating hormone (FSH) level > 35 mIU/mL.
    5. Women of child-bearing potential also include women who are using oral, implanted or injectable contraceptive hormones or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or where partner is sterile (eg, vasectomy), should be considered to be of child bearing potential.
21. ECOG Performance Status of 0-1
22. Age ≥ 18 years
23. Required Initial Laboratory Values:

    1. Granulocytes ≥ 1500 µL
    2. Hemoglobin ≥ 9.0 grams/dL (patient may be transfused to meet this criterion)
    3. Platelet count ≥ 100,000/µL
    4. Creatinine ≤ 1.5 x Upper limits of normal
    5. Bilirubin ≤ 1.5 mg/dL
    6. Albumin ≥ 2.5 g/dL
    7. Urinalysis ≤ 1 + protein*

       * *Patients discovered to have ≥ 2+ proteinuria at baseline must undergo a 24-hour urine collection that must demonstrate < 1 g of protein/24 hour or have a UPC < 1.0 to allow participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2334 (Actual)
Dates: Start 2005-11; Primary Completion 2015-02 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Venook, MD, Study Chair — University of California, San Francisco
Locations (683):
- United States (662):
  - Providence Cancer Center at Providence Hospital, Mobile, Alabama
  - Alaska Regional Hospital Cancer Center, Anchorage, Alaska
  - Providence Cancer Center, Anchorage, Alaska
  - Hembree Mercy Cancer Center at St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - NEA Medical Center - Stadium Boulevard, Jonesboro, Arkansas
  - Roy and Patricia Disney Family Cancer Center at Providence Saint Joseph Medical Center, Burbank, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Valley Medical Oncology Consultants - Castro Valley, Castro Valley, California
  - North Bay Cancer Center, Fairfield, California
  - Kaiser Permanente - Fremont, Fremont, California
  - Valley Medical Oncology, Fremont, California
  - Glendale Memorial Hospital Comprehensive Cancer Center, Glendale, California
  - California Cancer Care, Incorporated - Greenbrae, Greenbrae, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - Veterans Affairs Medical Center - Loma Linda (Pettis), Loma Linda, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Tibotec Therapeutics - Division of Ortho Biotech Products, LP, Marysville, California
  - Camino Medical Group - Treatment Center, Mountain View, California
  - El Camino Hospital Cancer Center, Mountain View, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons, Incorporated, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee, Incorporated, Oakland, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - St. Joseph Hospital Regional Cancer Center - Orange, Orange, California
  - Desert Regional Medical Center Comprehensive Cancer Center, Palm Springs, California
  - Palo Alto Medical Foundation, Palo Alto, California
  - Valley Medical Oncology Consultants - Pleasanton, Pleasanton, California
  - Kaiser Permanente Medical Center - Redwood City, Redwood City, California
  - Kaiser Permanente Medical Center - Richmond, Richmond, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - University of California Davis Cancer Center, Sacramento, California
  - South Sacramento Kaiser-Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Office -Vandever Medical Office, San Diego, California
  - Naval Medical Center - San Diego, San Diego, California
  - San Francisco General Hospital Medical Center, San Francisco, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Teresa, San Jose, California
  - Kaiser Foundation Hospital - San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Saint Helena Hospital, St. Helena, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - Tahoe Forest Cancer Center, Truckee, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - San Luis Valley Regional Medical Center, Alamosa, Colorado
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Memorial Hospital Cancer Center - Colorado Springs, Colorado Springs, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Kaiser Permanente - Denver, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Shaw Regional Cancer Center, Edwards, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Valley View Hospital Cancer Center, Glenwood Springs, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Kaiser Permanente - Lafayette, Lafayette, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Montrose Memorial Hospital Cancer Center, Montrose, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Bendheim Cancer Center at Greenwich Hospital, Greenwich, Connecticut
  - Helen and Harry Gray Cancer Center at Hartford Hospital, Hartford, Connecticut
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Middlesex Hospital Cancer Center, Middletown, Connecticut
  - George Bray Cancer Center at the Hospital of Central Connecticut - New Britain Campus, New Britain, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Kent General Hospital, Dover, Delaware
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Eugene M. and Christine E. Lynn Cancer Institute at Boca Raton Community Hospital - Main Campus, Boca Raton, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Lakeland Regional Cancer Center at Lakeland Regional Medical Center, Lakeland, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - Sacred Heart Medical Oncology, Pensacola, Florida
  - Phoebe Cancer Center at Phoebe Putney Memorial Hospital, Albany, Georgia
  - Northeast Georgia Cancer Care, LLC - Medical Oncology, Athens, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - John B. Amos Cancer Center, Columbus, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Dublin Hematology and Oncology Care, Dublin, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Cancer Center - Medical Oncology, Rome, Georgia
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Pearlman Comprehensive Cancer Center at South Georgia Medical Center, Valdosta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - Hawaii Medical Center - East, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kaiser Permanente - Moanalua Medical Center and Clinic, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Kauai Medical Clinic, Lihue, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute - Maui, Wailuku, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Creticos Cancer Center at Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Saint Joseph Hospital, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Sherman Hospital, Elgin, Illinois
  - Alexian Brothers Radiation Oncology, Elk Grove Village, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Evanston Hospital, Evanston, Illinois
  - St. Francis Hospital, Evanston, Illinois
  - Leonard C. Ferguson Cancer Center, Freeport, Illinois
  - Veterans Affairs Medical Center - Hines, Hines, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Provena St. Mary's Regional Cancer Center - Kankakee, Kankakee, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - Hematology Oncology Consultants - Naperville, Naperville, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Center for Cancer Care at OSF Saint Anthony Medical Center, Rockford, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Clarian Arnett Cancer Care, Lafayette, Indiana
  - Suniti Medical Corporation, Merrillville, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Community Hospital, Munster, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Heartland Oncology and Hematology, Council Bluffs, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Veterans Affairs Medical Center - Iowa City, Iowa City, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Covenant Cancer Treatment Center, Waterloo, Iowa
  - Hays Medical Center, Hays, Kansas
  - Hutchinson Hospital Corporation, Hutchinson, Kansas
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's Hospital - South, Overland Park, Kansas
  - Mount Carmel Regional Cancer Center, Pittsburg, Kansas
  - CCOP - Kansas City, Prairie Village, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - Ochsner Health Center - Bluebonnet, Baton Rouge, Louisiana
  - Ochsner Health Center - Covington, Covington, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - York Hospital's Oncology Treatment Center, York Village, Maine
  - DeCesaris Cancer Institute at Anne Arundel Medical Center, Annapolis, Maryland
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Veterans Affairs Medical Center - Baltimore, Baltimore, Maryland
  - National Naval Medical Center, Bethesda, Maryland
  - Shore Regional Cancer Center at Memorial Hospital - Easton, Easton, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Frederick Memorial Hospital Regional Cancer Therapy Center, Frederick, Maryland
  - John R. Marsh Cancer Center at Washington County Hospital, Hagerstown, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Caritas St. Elizabeth's Medical Center, Brighton, Massachusetts
  - Lahey Clinic Medical Center - Burlington, Burlington, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional Medical Center, Milford, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Caritas Norwood Hospital, Norwood, Massachusetts
  - NSMC Cancer Center - Peabody, Peabody, Massachusetts
  - Berkshire Hematology Oncology, PC, Pittsfield, Massachusetts
  - Commonwealth Hematology-Oncology, PC - Quincy, Quincy, Massachusetts
  - Baystate Regional Cancer Program at D'Amour Center for Cancer Care, Springfield, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Clemens Regional Medical Center, Mount Clemens, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - Michiana Hematology Oncology PC - Niles, Niles, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Alexandria, Minnesota
  - MeritCare Bemidji, Bemidji, Minnesota
  - St. Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - St. Luke's Hospital Cancer Care Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Keesler Air Force Base Medical Center, Keesler Air Force Base, Mississippi
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Central Care Cancer Center at Carrie J. Babb Cancer Center, Bolivar, Missouri
  - Skaggs Cancer Center at Skaggs Regional Medical Center, Branson, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Goldschmidt Cancer Center, Jefferson City, Missouri
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Parvin Radiation Oncology, Kansas City, Missouri
  - Heartland Hematology Oncology Associates, Incorporated, Kansas City, Missouri
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology, Incorporated, Saint Joseph, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Comprehensive Cancer Care, PC, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Saint Francis Cancer Treatment Center at Saint Francis Memorial Health Center, Grand Island, Nebraska
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - Callahan Cancer Center at Great Plains Regional Medical Center, North Platte, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Nevada Cancer Institute, Las Vegas, Nevada
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - Center for Cancer Care at Exeter Hospital, Exeter, New Hampshire
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Norris Cotton Cancer Center at Catholic Medical Center, Manchester, New Hampshire
  - Elliot Regional Cancer Center at Elliot Hospital, Manchester, New Hampshire
  - Oncology Center at St. Joseph Hospital, Nashua, New Hampshire
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - Dizzy Gillespie Cancer Institute at Englewood Hospital and Medical Center, Englewood, New Jersey
  - Hunterdon Regional Cancer Center at Hunterdon Medical Center, Flemington, New Jersey
  - CentraState Medical Center, Freehold, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Carol G. Simon Cancer Center at Morristown Memorial Hospital, Morristown, New Jersey
  - UMDNJ University Hospital, Newark, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Valley Hospital - Ridgewood, Ridgewood, New Jersey
  - Somerset Medical Center, Somerville, New Jersey
  - Frederick R. and Betty M. Smith Cancer Treatment Center, Sparta, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Falck Cancer Center at Arnot Ogden Medical Center, Elmira, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Tucker Center for Cancer Care at Orange Regional Medical Center, Middletown, New York
  - Winthrop University Hospital, Mineola, New York
  - Mount Kisco Medical Group, PC, Mount Kisco, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Interlakes Oncology/Hematology PC, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Nalitt Cancer Institute at Staten Island University Hospital, Staten Island, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Faxton Regional Cancer Center, Utica, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Alamance Cancer Center at Alamance Regional Medical Center, Burlington, North Carolina
  - Waverly Hematology Oncology, Cary, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Batte Cancer Center at Northeast Medical Center, Concord, North Carolina
  - CaroMont Cancer Center at Gaston Memorial Hospital, Gastonia, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - FirstHealth Moore Regional Community Hospital Comprehensive Cancer Center, Pinehurst, North Carolina
  - Rex Cancer Center at Rex Hospital, Raleigh, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - Nash Hospitals, Incorporated, Rocky Mount, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Marion L. Shepard Cancer Center at Beaufort County Hospital, Washington, North Carolina
  - Zimmer Cancer Center at New Hanover Regional Medical Center, Wilmington, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Roger Maris Cancer Center at MeritCare Hospital, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Trinity CancerCare Center, Minot, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Mercy Cancer Center at Mercy Medical Center, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel Hospital East, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - MedCentral - Mansfield Hospital, Mansfield, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Southern Ohio Medical Center Cancer Center, Portsmouth, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson Air Force Base, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma, LLC - Lawton, Lawton, Oklahoma
  - Cancer Care Associates - Norman, Norman, Oklahoma
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Cancer Care Associates - Mercy Campus, Oklahoma City, Oklahoma
  - Cancer Care Associates at Troy and Dollie Smith Cancer Center, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Willamette Falls Hospital, Oregon City, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Health Care - Portland, Portland, Oregon
  - Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Celilo Cancer Center at Mid-Columbia Medical Center, The Dalles, Oregon
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - St. Luke's Cancer Network at St. Luke's Hospital, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Doylestown Hospital Cancer Center, Doylestown, Pennsylvania
  - Delaware County Regional Cancer Center at Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Dale and Frances Hughes Cancer Center at Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Ephrata Cancer Center at Ephrata Community Hospital, Ephrata, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Riddle Memorial Hospital Cancer Center, Media, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Pottstown Memorial Regional Cancer Center, Pottstown, Pennsylvania
  - St. Joseph Medical Center, Reading, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Guthrie Cancer Center at Guthrie Clinic Sayre, Sayre, Pennsylvania
  - Hematology and Oncology Associates of Northeastern Pennsylvania, Scranton, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Associates in Hematology-Oncology, PC at Crozer Regional Cancer Center, Upland, Pennsylvania
  - Jennersville Regional Hospital, West Grove, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - Kent County Memorial Hospital, Warwick, Rhode Island
  - AnMed Cancer Center, Anderson, South Carolina
  - Keyserling Cancer Center at Beaufort Memorial Hospital, Beaufort, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - University of Tennessee Cancer Institute - Memphis, Memphis, Tennessee
  - MBCCOP - Meharry Medical College - Nashville, Nashville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Seton Shivers Cancer Program at Brackenridge Hospital, Austin, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - St. Luke's Texas Cancer Institute at St. Luke's Episcopal Hospital, Houston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - UMC Southwest Cancer and Research Center, Lubbock, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Virginia Oncology Associates - Hampton, Hampton, Virginia
  - Lynchburg Hematology-Oncology Clinic, Lynchburg, Virginia
  - Southwest Virginia Regional Cancer Center at Wellmonth Health, Norton, Virginia
  - Virginia Cancer Institute - West End, Richmond, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Island Hospital Cancer Care Center at Island Hospital, Anacortes, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Highline Medical Center Cancer Center, Burien, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center at Cabell Huntington Hospital, Huntington, West Virginia
  - Community Comprehensive Cancer Center at Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Princeton Community Hospital, Princeton, West Virginia
  - Langlade Memorial Hospital, Antigo, Wisconsin
  - Fox Valley Hematology and Oncology - East Grant Street, Appleton, Wisconsin
  - Marshfield Clinic - Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Vince Lombardi Cancer Clinic - Green Bay at Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercy Regional Cancer Center, Janesville, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Franciscan Skemp Healthcare - La Crosse Campus, La Crosse, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Dean Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Vince Lombardi Cancer Clinic - Marinette, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - D.N. Greenwald Center, Mukwonago, Wisconsin
  - Regional Cancer Center at Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - All Saints Cancer Center at Wheaton Franciscan Healthcare, Racine, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Saint Michael's Hospital Cancer Center, Stevens Point, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic - Two Rivers, Two Rivers, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
  - Marshfield Clinic - Wausau Center, Wausau, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
  - Oncology Alliance, SC - Milwaukee - West, Wauwatosa, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Riverview UW Cancer Center at Riverview Hospital, Wisconsin Rapids, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming
- Canada (21):
  - British Columbia Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Grand River Regional Cancer Centre at Grand River Hospital, Kitchener, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - R. S. McLaughlin Durham Regional Cancer Centre at Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
  - St. Catharines General Hospital at Niagara Health System, Saint Catharines, Ontario
  - Cancer Care Program at Thunder Bay Regional Health Sciences, Thunder Bay, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Odette Cancer Centre at Sunnybrook, Toronto, Ontario
  - St. Michael's Hospital - Toronto, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Trillium Health Centre - Mississauga Site, Toronto, Ontario
  - Windsor Regional Cancer Centre at Windsor Regional Hospital, Windsor, Ontario
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan

REFERENCES:
- [Background] Schrag D, Naughton M, Kesselheim A, et al.: Clinical trial participants' strategies for coping with prescription drug costs: A companion study to CALGB 80405. [Abstract] J Clin Oncol 27 (Suppl 15): A-9503, 2009.
- [Result] Venook AP, Blanke CD, Niedzwiecki D, Lenz HJ, Taylor JR, Hollis DR, Sutherland S, Goldberg RM. Revisiting the Cancer and Leukemia Group B/Southwest Oncology Group 80405 Trial: a phase III trial of chemotherapy and biologic agents for patients with untreated advanced colorectal adenocarcinoma. Clin Colorectal Cancer. 2007 May;6(7):536-8. doi: 10.3816/CCC.2007.n.021. No abstract available. PMID 17553204
- [Result] Venook AP, Blanke CD, Niedzwiecki D, Lenz HJ, Taylor JR, Hollis DR, Sutherland S, Goldberg RM. Cancer and Leukemia Group B/Southwest Oncology Group trial 80405: a phase III trial of chemotherapy and biologics for patients with untreated advanced colorectal adenocarcinoma. Clin Colorectal Cancer. 2005 Nov;5(4):292-4. doi: 10.3816/ccc.2005.n.043. No abstract available. PMID 16356309
- [Derived] Battaglin F, Ou FS, Qu X, Hochster HS, Niedzwiecki D, Goldberg RM, Mayer RJ, Ashouri K, Zemla TJ, Blanke CD, Venook AP, Kabbarah O, Lenz HJ, Innocenti F. HER2 Gene Expression Levels Are Predictive and Prognostic in Patients With Metastatic Colorectal Cancer Enrolled in CALGB/SWOG 80405. J Clin Oncol. 2024 Jun 1;42(16):1890-1902. doi: 10.1200/JCO.23.01507. Epub 2024 Mar 8. PMID 38457761
- [Derived] Raghav K, Ou FS, Venook AP, Innocenti F, Sun R, Lenz HJ, Kopetz S. Acquired Genomic Alterations on First-Line Chemotherapy With Cetuximab in Advanced Colorectal Cancer: Circulating Tumor DNA Analysis of the CALGB/SWOG-80405 Trial (Alliance). J Clin Oncol. 2023 Jan 20;41(3):472-478. doi: 10.1200/JCO.22.00365. Epub 2022 Sep 6. PMID 36067452
- [Derived] Yuan C, Sato K, Hollis BW, Zhang S, Niedzwiecki D, Ou FS, Chang IW, O'Neil BH, Innocenti F, Lenz HJ, Blanke CD, Goldberg RM, Venook AP, Mayer RJ, Fuchs CS, Meyerhardt JA, Ng K. Plasma 25-Hydroxyvitamin D Levels and Survival in Patients with Advanced or Metastatic Colorectal Cancer: Findings from CALGB/SWOG 80405 (Alliance). Clin Cancer Res. 2019 Dec 15;25(24):7497-7505. doi: 10.1158/1078-0432.CCR-19-0877. Epub 2019 Sep 23. PMID 31548349
- [Derived] Guercio BJ, Zhang S, Ou FS, Venook AP, Niedzwiecki D, Lenz HJ, Innocenti F, O'Neil BH, Shaw JE, Polite BN, Hochster HS, Atkins JN, Goldberg RM, Sato K, Ng K, Van Blarigan E, Mayer RJ, Blanke CD, O'Reilly EM, Fuchs CS, Meyerhardt JA. Associations of Physical Activity With Survival and Progression in Metastatic Colorectal Cancer: Results From Cancer and Leukemia Group B (Alliance)/SWOG 80405. J Clin Oncol. 2019 Oct 10;37(29):2620-2631. doi: 10.1200/JCO.19.01019. Epub 2019 Aug 13. PMID 31408415
- [Derived] Lenz HJ, Ou FS, Venook AP, Hochster HS, Niedzwiecki D, Goldberg RM, Mayer RJ, Bertagnolli MM, Blanke CD, Zemla T, Qu X, Wirapati P, Tejpar S, Innocenti F, Kabbarah O. Impact of Consensus Molecular Subtype on Survival in Patients With Metastatic Colorectal Cancer: Results From CALGB/SWOG 80405 (Alliance). J Clin Oncol. 2019 Aug 1;37(22):1876-1885. doi: 10.1200/JCO.18.02258. Epub 2019 May 1. PMID 31042420
- [Derived] Venook AP, Niedzwiecki D, Lenz HJ, Innocenti F, Fruth B, Meyerhardt JA, Schrag D, Greene C, O'Neil BH, Atkins JN, Berry S, Polite BN, O'Reilly EM, Goldberg RM, Hochster HS, Schilsky RL, Bertagnolli MM, El-Khoueiry AB, Watson P, Benson AB 3rd, Mulkerin DL, Mayer RJ, Blanke C. Effect of First-Line Chemotherapy Combined With Cetuximab or Bevacizumab on Overall Survival in Patients With KRAS Wild-Type Advanced or Metastatic Colorectal Cancer: A Randomized Clinical Trial. JAMA. 2017 Jun 20;317(23):2392-2401. doi: 10.1001/jama.2017.7105. PMID 28632865
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: From 5/2005 to 9/2009, patients were randomized 1:1:1 to Arms A, B and C. Study was amended in 2009 to include only KRAS wild type patients; then Arm C was closed based on data showing no benefit from chemo with the combination of Bevacizumab and an EGFR antibody. Thereafter, only KRAS wild type patients were randomized 1:1 to Arm A and B.
Period: Overall Study
Arm/Group | Arm A: FOLFOX or FOLFIRI + Bevacizumab | Arm B: FOLFOX or FOLFIRI + Cetuximab | Arm C: FOLFOX or FOLFIRI + Cetuximab + Bevacizumab
Started | 899 | 902 | 533
Completed | 899 | 902 | 533
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: During the trial, it was learned that KRAS mutation predicted for lack of efficacy of EGFR antibodies; also studies showed no benefit from chemo combined with both Bevacizumab and an EGFR antibody. The trial was amended to 2 arms limited to KRAS wild type patients. Only confirmed and consented KRAS wild type patients were analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: FOLFOX or FOLFIRI + Bevacizumab | Arm B: FOLFOX or FOLFIRI + Cetuximab | Arm C: FOLFOX or FOLFIRI + Cetuximab + Bevacizumab | Total
Number analyzed (Participants) | 559 | 578 | 0 | 1137
Age, Continuous [Median (Full Range); unit: years] | 59 [21.8 to 85] | 59.2 [20.8 to 89.5] |  | 59.1 [20.8 to 89.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 211 | 229 |  | 440
  Male | 348 | 349 |  | 697
Region of Enrollment [Number; unit: participants]
  Canada | 32 | 32 |  | 64
  United States | 527 | 546 |  | 1073

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Survival time will be defined as the time from registration to death. Time to event distributions will be estimated using the Kaplan-Meier method. Overall Survival (OS) will be compared between Arm A and Arm B.
Time Frame: Up to 5 years post-treatment
Population: All eligible KRAS wild type patients that began treatment were included in this endpoint.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: FOLFOX or FOLFIRI + Bevacizumab | Arm B: FOLFOX or FOLFIRI + Cetuximab | Arm C: FOLFOX or FOLFIRI + Cetuximab + Bevacizumab
Number analyzed (Participants) | 559 | 578 | 0
months | 29.0 [25.6 to 31.2] | 30.0 [27.5 to 32.8] |
Statistical Analysis 1: Comparison: Arm A: FOLFOX or FOLFIRI + Bevacizumab vs Arm B: FOLFOX or FOLFIRI + Cetuximab; Test type: Superiority; p = 0.08, Log Rank; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.77 to 1.01]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS will be measured from study entry until first documented progression or death from any cause. Time to event distributions will be estimated using the Kaplan-Meier method. PFS will be compared between Arm A and Arm B.
Time Frame: Up to 5 years post-treatment
Population: All eligible KRAS wild type patients were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: FOLFOX or FOLFIRI + Bevacizumab | Arm B: FOLFOX or FOLFIRI + Cetuximab | Arm C: FOLFOX or FOLFIRI + Cetuximab + Bevacizumab
Number analyzed (Participants) | 559 | 578 | 0
months | 10.6 [9.5 to 11.1] | 10.5 [9.5 to 11.3] |
Statistical Analysis 1: Comparison: Arm A: FOLFOX or FOLFIRI + Bevacizumab vs Arm B: FOLFOX or FOLFIRI + Cetuximab; Test type: Superiority; p = 0.45, Log Rank; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.84 to 1.08]

3. Secondary Outcome: Time to Treatment Failure
Time Frame: Up to 5 years post-treatment
Reporting Status: Not Posted

4. Secondary Outcome: Duration of Tumor Response
Time Frame: Up to 5 years post-treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Analysis was conducted on all KRAS wild type patients that were treated and assessed for adverse events.
Arm/Group | Arm A: FOLFOX or FOLFIRI + Bevacizumab | Arm B: FOLFOX or FOLFIRI + Cetuximab
Serious Adverse Events (participants affected / at risk) | 98/559 | 111/578
Other Adverse Events (participants affected / at risk) | 531/559 | 548/578
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: FOLFOX or FOLFIRI + Bevacizumab (N=559) | Arm B: FOLFOX or FOLFIRI + Cetuximab (N=578)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 3 (3) | 1 (1)
Eye disorder (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 3 (3)
Colonic perforation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Jejunal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death NOS (General disorders) | 5 (5) | 2 (2)
Disease progression (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 4 (4) | 3 (3)
Sudden death (General disorders) | 2 (2) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Ileal infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 4 (4)
Arterial injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 2 (3) | 7 (9)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Carbon monoxide diffusing capacity decreased (Investigations) | 0 (0) | 2 (2)
Cardiac troponin I increased (Investigations) | 2 (2) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Leukocyte count decreased (Investigations) | 2 (2) | 2 (2)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 35 (38) | 36 (43)
Platelet count decreased (Investigations) | 2 (2) | 3 (3)
Serum cholesterol increased (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1) | 4 (5)
Blood uric acid increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 0 (0) | 5 (12)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum sodium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 2 (2) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Thrombosis (Vascular disorders) | 14 (14) | 22 (39)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: FOLFOX or FOLFIRI + Bevacizumab (N=559) | Arm B: FOLFOX or FOLFIRI + Cetuximab (N=578)
Blood disorder (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 10 (10)
Hemoglobin decreased (Blood and lymphatic system disorders) | 95 (161) | 83 (145)
Hemolysis (Blood and lymphatic system disorders) | 7 (7) | 5 (6)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphatic disorder (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 5 (5)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 5 (5) | 1 (1)
Cardiac pain (Cardiac disorders) | 4 (4) | 5 (5)
Conduction disorder (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 2 (2) | 3 (6)
Myocardial ischemia (Cardiac disorders) | 3 (3) | 5 (5)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Nodal arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 3 (3)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 5 (5)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Ventricular trigeminy (Cardiac disorders) | 1 (1) | 1 (1)
Ear disorder (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (2) | 1 (1)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Hearing test abnormal (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 4 (5) | 4 (7)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Cushingoid (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (2) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (2) | 1 (1)
Cataract (Eye disorders) | 3 (3) | 1 (3)
Conjunctivitis (Eye disorders) | 3 (4) | 12 (23)
Diplopia (Eye disorders) | 1 (1) | 1 (1)
Dry eye syndrome (Eye disorders) | 1 (1) | 1 (3)
Extraocular muscle paresis (Eye disorders) | 0 (0) | 1 (2)
Eye disorder (Eye disorders) | 0 (0) | 4 (7)
Eye pain (Eye disorders) | 1 (1) | 1 (1)
Eyelid function disorder (Eye disorders) | 0 (0) | 2 (6)
Glaucoma (Eye disorders) | 0 (0) | 1 (2)
Keratitis (Eye disorders) | 0 (0) | 1 (1)
Retinopathy (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 3 (5) | 2 (10)
Watering eyes (Eye disorders) | 1 (1) | 4 (8)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 189 (377) | 186 (327)
Anal exam abnormal (Gastrointestinal disorders) | 2 (2) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (2) | 0 (0)
Anal hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anal mucositis (Gastrointestinal disorders) | 0 (0) | 1 (3)
Anal pain (Gastrointestinal disorders) | 3 (5) | 3 (6)
Ascites (Gastrointestinal disorders) | 3 (3) | 2 (2)
Cheilitis (Gastrointestinal disorders) | 2 (3) | 5 (5)
Colitis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Colonic fistula (Gastrointestinal disorders) | 2 (5) | 1 (1)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 5 (5) | 6 (6)
Colonic perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 41 (57) | 58 (91)
Diarrhea (Gastrointestinal disorders) | 304 (751) | 346 (804)
Dry mouth (Gastrointestinal disorders) | 1 (2) | 7 (10)
Duodenal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 23 (27) | 19 (57)
Dysphagia (Gastrointestinal disorders) | 9 (9) | 6 (6)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 21 (28) | 54 (71)
Endoscopy small intestine abnormal (Gastrointestinal disorders) | 1 (1) | 1 (3)
Enteritis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Esophageal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 3 (5) | 4 (4)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 2 (2)
Fistula of small intestine (Gastrointestinal disorders) | 2 (3) | 0 (0)
Flatulence (Gastrointestinal disorders) | 6 (11) | 11 (12)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 4 (7) | 6 (25)
Gastrointestinal disorder (Gastrointestinal disorders) | 6 (11) | 8 (9)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 12 (18) | 13 (16)
Ileal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 6 (8) | 1 (1)
Intestinal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Jejunal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 44 (57) | 59 (102)
Nausea (Gastrointestinal disorders) | 90 (114) | 100 (154)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 2 (3) | 4 (5)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Periodontal disease (Gastrointestinal disorders) | 1 (3) | 2 (6)
Peritoneal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 5 (6) | 3 (3)
Rectal mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 15 (27) | 7 (12)
Rectal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (2)
Salivary gland disorder (Gastrointestinal disorders) | 2 (4) | 0 (0)
Small intestinal mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 7 (7) | 7 (7)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestine ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 2 (4)
Tooth disorder (Gastrointestinal disorders) | 1 (2) | 4 (4)
Toothache (Gastrointestinal disorders) | 4 (4) | 3 (3)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 174 (284) | 185 (265)
Chest pain (General disorders) | 11 (15) | 7 (7)
Chills (General disorders) | 43 (51) | 62 (88)
Edema limbs (General disorders) | 7 (7) | 9 (15)
Facial pain (General disorders) | 1 (1) | 5 (5)
Fatigue (General disorders) | 397 (1213) | 418 (1315)
Fever (General disorders) | 75 (101) | 67 (83)
Flu-like symptoms (General disorders) | 0 (0) | 2 (2)
Gait abnormal (General disorders) | 1 (1) | 1 (1)
General symptom (General disorders) | 6 (7) | 5 (8)
Injection site reaction (General disorders) | 2 (3) | 3 (3)
Localized edema (General disorders) | 2 (3) | 1 (1)
Pain (General disorders) | 28 (39) | 30 (32)
Pericardial pain (General disorders) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Gallbladder pain (Hepatobiliary disorders) | 1 (2) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatobiliary disease (Hepatobiliary disorders) | 2 (2) | 0 (0)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 3 (3)
Cytokine release syndrome (Immune system disorders) | 22 (29) | 56 (61)
Hypersensitivity (Immune system disorders) | 13 (14) | 15 (20)
Abdominal infection (Infections and infestations) | 2 (2) | 0 (0)
Anal infection (Infections and infestations) | 1 (3) | 2 (3)
Anorectal infection (Infections and infestations) | 2 (2) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 10 (14) | 7 (8)
Bone infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 4 (7) | 1 (1)
Catheter related infection (Infections and infestations) | 14 (17) | 10 (10)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1) | 1 (1)
Conjunctivitis infective (Infections and infestations) | 1 (1) | 6 (7)
Device related infection (Infections and infestations) | 1 (1) | 2 (2)
Esophageal infection (Infections and infestations) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 2 (2) | 2 (5)
Gingival infection (Infections and infestations) | 5 (6) | 0 (0)
Infection (Infections and infestations) | 16 (19) | 17 (22)
Infection with unknown ANC (Infections and infestations) | 0 (0) | 1 (1)
Infection without neutropenia (Infections and infestations) | 2 (2) | 2 (3)
Infectious colitis (Infections and infestations) | 1 (1) | 3 (3)
Infectious meningitis (Infections and infestations) | 0 (0) | 1 (1)
Joint infection (Infections and infestations) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Lip infection (Infections and infestations) | 2 (2) | 2 (2)
Lymph gland infection (Infections and infestations) | 0 (0) | 1 (1)
Mediastinal infection (Infections and infestations) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 2 (2)
Nail infection (Infections and infestations) | 0 (0) | 16 (30)
Opportunistic infection (Infections and infestations) | 3 (3) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (2)
Otitis media (Infections and infestations) | 3 (3) | 1 (1)
Paranasal sinus infection (Infections and infestations) | 1 (2) | 0 (0)
Pelvic infection (Infections and infestations) | 1 (1) | 0 (0)
Penile infection (Infections and infestations) | 0 (0) | 1 (1)
Peripheral nerve infection (Infections and infestations) | 1 (1) | 0 (0)
Peritoneal infection (Infections and infestations) | 3 (3) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 7 (7) | 8 (10)
Rhinitis infective (Infections and infestations) | 2 (2) | 1 (1)
Salivary gland infection (Infections and infestations) | 0 (0) | 1 (1)
Scrotal infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 5 (5)
Sinusitis (Infections and infestations) | 7 (9) | 3 (4)
Skin infection (Infections and infestations) | 5 (6) | 19 (24)
Small intestine infection (Infections and infestations) | 1 (1) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 1 (1)
Stoma site infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 8 (11) | 4 (5)
Upper aerodigestive tract infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 10 (16) | 7 (9)
Urethral infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 24 (27) | 19 (21)
Vaginal infection (Infections and infestations) | 3 (4) | 0 (0)
Wound infection (Infections and infestations) | 4 (5) | 6 (7)
Wound-infectious (Infections and infestations) | 0 (0) | 1 (1)
Aortic injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Esophageal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 3 (3) | 5 (6)
Intestinal stoma site bleeding (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Intraoperative gastrointestinal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 0 (0) | 5 (5)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 14 (24) | 21 (33)
Wound dehiscence (Injury, poisoning and procedural complications) | 5 (7) | 1 (2)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 3 (3)
Alanine aminotransferase increased (Investigations) | 16 (29) | 23 (38)
Alkaline phosphatase (Investigations) | 1 (1) | 1 (1)
Alkaline phosphatase increased (Investigations) | 32 (49) | 35 (58)
Amylase increased (Investigations) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 11 (15) | 21 (34)
Blood bilirubin increased (Investigations) | 45 (84) | 57 (108)
Blood gonadotrophin abnormal (Investigations) | 1 (2) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 1 (4)
Cardiac troponin T increased (Investigations) | 0 (0) | 1 (1)
Coagulopathy (Investigations) | 0 (0) | 2 (6)
Creatinine increased (Investigations) | 21 (25) | 7 (8)
Electrocardiogram QTc interval prolonged (Investigations) | 0 (0) | 1 (1)
Fibrinogen decreased (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 4 (9)
INR increased (Investigations) | 10 (14) | 18 (40)
Laboratory test abnormal (Investigations) | 2 (2) | 7 (8)
Leukocyte count decreased (Investigations) | 79 (144) | 98 (150)
Lipase increased (Investigations) | 1 (1) | 4 (4)
Lymphocyte count decreased (Investigations) | 29 (68) | 31 (60)
Neutrophil count decreased (Investigations) | 316 (716) | 334 (792)
Platelet count decreased (Investigations) | 208 (541) | 210 (575)
Serum cholesterol increased (Investigations) | 1 (2) | 3 (11)
Weight gain (Investigations) | 10 (30) | 9 (21)
Weight loss (Investigations) | 35 (49) | 63 (113)
Anorexia (Metabolism and nutrition disorders) | 71 (92) | 100 (142)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Blood glucose increased (Metabolism and nutrition disorders) | 75 (141) | 80 (161)
Dehydration (Metabolism and nutrition disorders) | 53 (62) | 53 (66)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1) | 2 (4)
Serum albumin decreased (Metabolism and nutrition disorders) | 64 (87) | 62 (90)
Serum calcium decreased (Metabolism and nutrition disorders) | 25 (26) | 36 (51)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Serum glucose decreased (Metabolism and nutrition disorders) | 5 (7) | 5 (6)
Serum magnesium decreased (Metabolism and nutrition disorders) | 56 (97) | 231 (685)
Serum magnesium increased (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 10 (14) | 25 (35)
Serum potassium decreased (Metabolism and nutrition disorders) | 29 (37) | 56 (72)
Serum potassium increased (Metabolism and nutrition disorders) | 4 (4) | 10 (11)
Serum sodium decreased (Metabolism and nutrition disorders) | 16 (24) | 10 (11)
Serum sodium increased (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Serum triglycerides increased (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 27 (56) | 14 (18)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 29 (56) | 29 (45)
Bone pain (Musculoskeletal and connective tissue disorders) | 6 (12) | 9 (13)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Joint disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 15 (17)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 4 (5) | 4 (5)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (12) | 11 (17)
Neck pain (Musculoskeletal and connective tissue disorders) | 5 (7) | 4 (4)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 (36) | 21 (28)
Soft tissue necrosis upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Upper extremity dysfunction (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (7)
Ataxia (Nervous system disorders) | 3 (3) | 7 (10)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 4 (4) | 2 (2)
Dizziness (Nervous system disorders) | 19 (25) | 28 (31)
Dysgeusia (Nervous system disorders) | 24 (37) | 33 (47)
Extrapyramidal disorder (Nervous system disorders) | 2 (2) | 2 (11)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 98 (209) | 80 (165)
Ischemia cerebrovascular (Nervous system disorders) | 2 (2) | 4 (4)
Memory impairment (Nervous system disorders) | 1 (1) | 2 (2)
Mini mental status examination abnormal (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (2) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 5 (5) | 3 (3)
Peripheral motor neuropathy (Nervous system disorders) | 9 (33) | 12 (20)
Peripheral sensory neuropathy (Nervous system disorders) | 355 (1131) | 344 (1176)
Recurrent laryngeal nerve palsy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 5 (5)
Sinus pain (Nervous system disorders) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 5 (7) | 3 (4)
Syncope (Nervous system disorders) | 10 (10) | 17 (19)
Syncope vasovagal (Nervous system disorders) | 1 (1) | 2 (2)
Tremor (Nervous system disorders) | 1 (1) | 3 (5)
Trigeminal nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 3 (3)
Anxiety (Psychiatric disorders) | 22 (47) | 12 (18)
Confusion (Psychiatric disorders) | 6 (6) | 5 (5)
Depression (Psychiatric disorders) | 16 (19) | 23 (36)
Insomnia (Psychiatric disorders) | 26 (34) | 36 (65)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Bladder hemorrhage (Renal and urinary disorders) | 2 (2) | 1 (1)
Bladder pain (Renal and urinary disorders) | 0 (0) | 2 (2)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis (Renal and urinary disorders) | 0 (0) | 3 (3)
Glomerular filtration rate decreased (Renal and urinary disorders) | 0 (0) | 2 (2)
Hemoglobin urine positive (Renal and urinary disorders) | 2 (3) | 0 (0)
Hemorrhage urinary tract (Renal and urinary disorders) | 2 (3) | 2 (2)
Kidney pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Kidney perforation (Renal and urinary disorders) | 1 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 159 (335) | 43 (62)
Renal failure (Renal and urinary disorders) | 7 (7) | 3 (3)
Renal hemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteric hemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 2 (7)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 6 (8) | 4 (4)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 5 (9)
Urinary retention (Renal and urinary disorders) | 5 (8) | 2 (3)
Urogenital disorder (Renal and urinary disorders) | 1 (1) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 2 (3) | 1 (4)
Gynecomastia (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 2 (3) | 3 (4)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (3) | 1 (1)
Vaginal mucositis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 9 (16) | 4 (4)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (21) | 11 (29)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 33 (53) | 37 (61)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (9) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 18 (29) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 4 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 8 (8)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (4)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 9 (9)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tracheoscopy abnormal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 4 (12) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 16 (35) | 18 (27)
Body odor (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (12) | 38 (74)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 (3) | 11 (18)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 24 (53) | 46 (71)
Nail disorder (Skin and subcutaneous tissue disorders) | 6 (8) | 20 (40)
Pain of skin (Skin and subcutaneous tissue disorders) | 2 (2) | 7 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 23 (27)
Rash acneiform (Skin and subcutaneous tissue disorders) | 9 (15) | 123 (271)
Rash desquamating (Skin and subcutaneous tissue disorders) | 13 (16) | 66 (110)
Rash/dermatitis associated with high-dose chemotherapy or BMT studies. (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 5 (6) | 31 (53)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 6 (15) | 6 (16)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5)
Sweating (Skin and subcutaneous tissue disorders) | 9 (12) | 7 (21)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1) | 4 (8)
Hypertension (Vascular disorders) | 179 (402) | 80 (184)
Hypotension (Vascular disorders) | 23 (25) | 35 (40)
Lymph leakage (Vascular disorders) | 1 (1) | 0 (0)
Lymphedema (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 2 (3) | 2 (2)
Thrombosis (Vascular disorders) | 44 (97) | 50 (95)
Vascular disorder (Vascular disorders) | 2 (2) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less